# **Emotion Focused Therapy for Competitive Athletes**

Please read the information letter and consent form below.

| 1) | Date and Time: | |
|----|----------------|-------------|
| | | <del></del> |



 $\mathbf{REDCap}^{\circ}$ 

## Emotion Focused Therapy for Competitive Athletes

#### Contact Information

Primary Investigators:
Dr. Katherine Tamminen, Associate Professor University of Toronto
Faculty of Kinesiology & Physical Education
55 Harbord Street, Toronto, ON, M5S 2W6 katherine.Tamminen@utoronto.ca
(416) 946-4068

Dr. Jeanne Watson, Professor University of Toronto Ontario Institute for Studies in Education 252 Bloor Street West, Toronto, ON, M5S 1V6 jeanne.watson@utoronto.ca (416) 978-0705

Research Assistants/Student Therapists: J'mi Worthen jmi.worthen@mail.utoronto.ca

Susan Osher susan.osher@mail.utoronto.ca

Yehuda Gabler yehuda.gabler@mail.utoronto.ca

## Information Letter

## Study Overview:

The purpose of this pilot study is to examine the use of Emotion Focused Therapy among competitive athletes over the age of 18 in Ontario. Emotion Focused Therapy is an approach to psychotherapy that focuses on emotions to address concerns such as depression, and anxiety. Emotion Focused Therapy promotes emotional awareness and understanding, emotional expression, and emotion regulation. It is an evidence-based approach to psychotherapy that has been used to treat issues such as depression and anxiety in the general population; however, it has not been tested specifically with competitive athletes. The purpose of this study is to evaluate the use of Emotion Focused Therapy for athletes experiencing mild to moderate depression and/or anxiety.

For more information about Emotion Focused Therapy, please see the following links:

What is Emotion Focused Therapy - International Society for Emotion Focused Therapy

Emotion Focused Therapy - goodtherapy.org

## What is involved?

If you agree to participate, you will be asked to complete a screening survey to determine your eligibility to take part in this study. The survey will ask for demographic information, as well as questions about your emotions, sport experiences, and symptoms of anxiety and depression. Your responses will be screened by a research coordinator who will contact you about your scores and to determine whether the intervention will be a good fit for you.

If you are eligible to participate in the study, you will be assigned to receive 12 weekly sessions of Emotion Focused Therapy with a trained student therapist. Each session will be held individually and will be 1 hour long. Each session will be held online via Microsoft Teams and the sessions will be video recorded.

03/25/2023 5:14pm projectredcap.org

You may be assigned to start the therapy immediately, or you may be required to wait up to 12 weeks before you can begin the therapy sessions. If you are assigned to wait before beginning therapy, you will be asked not to seek additional or alternative therapy or treatment while you are waiting. However, if your symptoms worsen or you are in need of immediate psychological support, please contact Crisis Services Canada (1-833-456-4566) or visit http://www.crisisservicescanada.ca/en/ If you are in immediate distress, call 911.

During the study, you will be asked to complete three additional surveys. Each survey is expected to take 30-45min to complete.

At the end of the study, you will also be asked to participate in an interview. The interview will last approximately 30-45min and you will be asked questions about your experience during the study. For example, you will be asked about the therapy you received, benefits or difficulties you experienced during the study, and recommendations for future interventions with athletes.

If you have any concerns about your mental health please contact the support services provided at the end of this information letter.

## Who can participate?

Competitive athletes - competitive means the primary focus in your sport is on performance improvement and competition in a specific sport, typically training more than 3 times per week, competing at the provincial level or higher (for example: varsity or collegiate athletes, athletes competing provincially, nationally, or internationally) Over the age of 18 Living in Ontario Experiencing mild to moderate depression and/or anxiety Not currently receiving therapy for depression/anxiety Interested individuals can complete the screening measures on the next page to determine your eligibility to participate.

#### What are the benefits?

Athletes may benefit from taking part in this study and receiving 12 individual psychotherapy sessions with a trained student therapist at no cost. Other studies have demonstrated that Emotion Focused Therapy is an effective approach for helping people experiencing symptoms of depression and anxiety, and athletes may benefit by experiencing an improvement in depression or anxiety symptoms.

The results from this study will also help expand the field of sports psychology and provide information about the use of Emotion Focused Therapy among competitive athletes.

Athletes who complete the study will be eligible to receive \$25 for each survey they complete. Athletes will also be eligible to receive \$25 for participating in the interview at the end of the study. If you stop participating in the study (i.e., stop the therapy sessions and do not complete the remaining surveys), you will be compensated for the surveys that you have completed to that point. The compensation will be provided at the end of study.

## Are there any risks?

Although Emotion Focused Therapy has been shown to help people with symptoms of depression and anxiety, there is a possibility that it may not help you. It is also not uncommon for people to experience an increase in symptoms or emotional discomfort before experiencing improvement. If you experience worsening symptoms and require immediate support while you are participating in the study, you can contact emergency psychological support sevices: Crisis Services Canada (1-833-456-4566) or visit http://www.crisisservicescanada.ca/en/ If you are in immediate distress, call 911.

Answering questions about your emotions, well-being, and mental health might make you feel uncomfortable or upset. To reduce this risk, you can stop completing the questionnaire at any point, and you can withdraw from the study at any time.

Some survey questions may ask about risk of self-harm or suicide intentions. Responses to these questions will be screened by a research coordinator. If there are concerns about your immediate safety, we will contact you within 24 hours to provide emergency mental health support services.

If you feel the need to access help or would like to further discuss any feelings or concerns, please refer to the list of support services included below.

Survey Data. All electronic data will be held on a password protected, encrypted computer in the Sport and Performance Psychology Lab at the University of Toronto in the Faculty of Kinesiology and Physical Education (room 425B, Goldring Centre for High Performance Sport). The surveys are online, so there will be no paper records. Only the researchers will have access to the information you provide, and your identifying information (email and phone number) will be removed from the dataset and your responses will be assigned a participant number.

Once the study is complete, the anonymous survey data will be stored indefinitely as a password-protected file on an online database (Dataverse) for future research analysis. The survey data is not publicly available, and future researchers will be required to obtain ethical approval to access the dataset. No names or identifying information will be stored for future research.

Interview Data. If you choose to take part in an interview at the end of the study, the interview will be video recorded and then transcribed. After the interview is transcribed, the video will be permanently deleted. The transcript will be de-identified and personally identifying information will be removed from the transcripts. The transcripts will be stored on a secure computer server at the University of Toronto and will only be accessible to the research team.

Once the study is complete, the results will be presented at a conference and published in an academic journal. The information you provide will only be used for research purposes, and your name, sport, and any identifying information will not be linked with your data. Only general information will be reported (e.g., "25% of athletes reported experiencing symptoms of anxiety"). A summary of the research results will be sent to all study participants at the end of the study.

Therapy Sessions. The video recorded therapy sessions will be saved in a password-protected folder on a secure computer server in the Faculty of Kinesiology and Physical Education. The video recordings will be saved indefinitely for future analysis and training purposes. For example, future research analysis may include examining the types of issues discussed in the therapy sessions, or an examination of the interactions between the student therapist and the participants. The videos will not be stored on a public database; they will only be stored on the University of Toronto's computer servers. In the future if researchers wish to access this data, they must have ethical approval and demonstrate appropriate training in psychotherapy research approaches. Researchers wishing to use the data for research purposes would have to contact Dr. Tamminen with a request to access the data, and they must have ethical approval by their research ethics board.

Mandatory Reporting and Limits to Confidentiality. Although your information will be kept confidential, there are some situations where we are unable to maintain confidentiality. During the therapy sessions, if you experience symptoms of distress, or if the therapist has grounds to believe there is a risk of harm to yourself or others, the therapist will contact emergency services to ensure your safety. The therapist is also required to inform appropriate authorities if there is a risk of harm to a child in need of protection, or if an individual in a long term care home is at risk of harm. Finally, if you tell the therapist that you have experienced sexual abuse by a regulated health professional (e.g., a doctor, etc.), that must also be reported to the appropriate authorities.

## Freedom to Withdraw

Participation in this study is voluntary. There will be no negative consequences if you do not participate, and we will not tell your coach or anyone else about who chooses to participate or not participate in the study. If you do not want to participate in this study, it will not impact your position/reputation/relationship with the team.

You can choose to stop participating in the study at any time by ending the survey (e.g., closing the internet browser window), or by stopping your participation in the therapy sessions. If you decide to stop participating in the study, you may be contacted by the therapist or by the research coordinator to ensure your safety and to ask if you need any additional support or services.

If you stop participating in the study before completing the survey and would like to remove your data from the study, you may contact Katherine Tamminen to ask for your data to be removed. You may contact us up until June 30, 2024 to remove your data from the study; after this point the analysis will be completed and it will not be possible to remove your data from the study.

If you have questions about this study, or about the information used for research purposes, you may contact Dr. Katherine Tamminen (katherine.tamminen@utoronto.ca). You may also contact the Research Oversight and Compliance Office - Human Research Ethics Program at ethics.review@utoronto.ca or 416-946-3273 if you have questions about your rights as a participant in this study. The research study you are participating in may be reviewed for quality assurance to make sure that the required laws and guidelines are followed. If chosen, (a) representative(s) of the Human Research Ethics Program (HREP) may access study-related data and/or consent materials as part of the review. All information accessed by the HREP will be upheld to the same level of confidentiality that has been stated by the research team.

List of Support Services

Canadian Mental Health Association - Regional Office Phone Numbers:

Alberta: (780) 482-6576

British Columbia: (604) 688-3234

Manitoba: 204-982-6100

New Brunswick: (506) 455-5231

Newfoundland and Labrador: (709) 753-8550

Northwest Territories: (867) 873-3190

Nova Scotia: (902) 466-6600

Nunavut Kamatsiagtut Help Line: 1-867-979-3333

Ontario Division: (416) 977-5580

Prince Edward Island: (902) 566-3034

Quebec: (514) 521-4993

Saskatchewan: 306-525-5601

Yukon: (867) 668-6429

For more information, please visit: https://cmha.ca/

Athletes can also contact the Canadian Centre for Mental Health and Sport at: https://www.ccmhs-ccsms.ca/

## Consent of Participant

To complete the screening measures and determine your eligibility for the study, please read the information below.

By checking "yes" below, I indicate that:

- 1. I understand that I have been asked to participate in a study to test the use of Emotion Focused Therapy among competitive athletes.
- 2. I understand the benefits and risks involved in taking part in this study.
- 3. I understand that I may be asked to wait up to 12 weeks before beginning therapy for this study. During this time, I will not seek other therapy unless my symptoms worsen and I am in need of immediate psychological support.
- 4. I understand that if I have questions, I may contact Katherine Tamminen (primary investigator) or Jeffrey Zeuner (research coordinator) about this survey.
- 5. I understand that my answers on the survey will be used for research purposes.
- 6. I understand that the therapy sessions will be held online using Microsoft Teams and the sessions will be video recorded.
- 7. I understand that only the members of the research team will have access to my data during the study.
- 8. I understand that participating in this study or withdrawing from this study will not have any negative consequences for me as an athlete.
- 9. I understand that I can contact the researchers if I want to remove my data from the study.
- 10. I understand that my data (with all identifying information removed) will be stored indefinitely on an online database for future research purposes, and future researchers will need ethical approval to access the data.

| <b>Z</b> ) | r consent to participate in this study: | ○ No |
|------------|-----------------------------------------|------|
| 3) | Email: | |
| 4) | Phone: | |

